CLINICAL TRIAL: NCT03897998
Title: Neural Correlates of Hypoalgesia Driven by Observation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Luana Colloca, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00085382
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pain; Virtual Reality; Placebo
Keywords: Naloxone; fMRI; EEG; Observation; Healthy Volunteers
MeSH Terms: conditions — Pain | interventions — Naloxone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This will be a 2 (group: naloxone vs. saline) X 2 (condition: placebo vs. control) double-blind mixed experimental design with group as the between-subjects factor and condition as the within-subjects factor. Each participant will be randomly assigned to either the naloxone or the saline group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The UM Pharmacy will assign de-identified study IDs to participants and provide the study drug (Naloxone or Saline) so that participants, the person conducting the experiment, and the investigator will be blind to the participant's group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naloxone (Active Comparator): NARCAN® Naloxone Nasal Spray will be used to block placebo effects during the fMRI experiment. Participants will be stratified for sex and then randomized to naloxone (The dose of naloxone will be 4 mg, so 0.1 mL of 40 mg/ml naloxone solution given intranasally) or saline (0.1 mL 0.9% sodium chloride intranasally), respectively. Investigators, staff, and participants will be blinded to the treatment options.
  Interventions: Drug: Naloxone
- Saline (Sham Comparator): Saline will be used as a sham comparator for blocking placebo effects during the fMRI experiment. Participants will be stratified for sex and then randomized to naloxone (The dose of naloxone will be 4 mg, so 0.1 mL of 40 mg/ml naloxone solution given intranasally) or saline (0.1 mL 0.9% sodium chloride intranasally), respectively. Investigators, staff, and participants will be blinded to the treatment options.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Naloxone — 4mg of Naloxone will be administered (0.1 mL of 40 mg/ml naloxone solution given intranasally).
  A random allocation sequence will be independently generated by the UM Pharmacy. The Principal investigator will call for each experiment.
  Other Names: Naloxone Hydrochloride/Narcan Intranasal
  Arms: Naloxone
Other: Saline — Intranasal Normal Saline (0.1 mL 0.9% sodium chloride) will be administered shortly before beginning the fMRI experiment.
  A random allocation sequence will be independently generated by the UM Pharmacy. The Principal investigator will call for each experiment.
  Other Names: Sodium chloride
  Arms: Saline

SUMMARY:
Placebo effects held an ambivalent place in health care for at least two centuries. On the one hand, placebos are traditionally used as controls in clinical trials to correct for biases and the placebo response is viewed as an effect to be factored out in order to isolate and accurately measure the effects of the treatment. On the other hand, there is scientific evidence that placebo effects represent fascinating psychoneurobiological events involving the contribution of distinct central nervous as well as peripheral physiological mechanisms that influence pain perception and clinical pain symptoms and substantially modulate the response to pain therapeutics. Therefore, placebo effects have shifted from being a challenge for clinical trials to a resource to trigger the reduction of pain based on endogenous mechanisms that can be activated in the brain to promote hypolagesia, self-healing, and well-being. This is relevant in acute pain settings given that chronic opioid users die within approximately 2.5 years of being prescribed their first opioid medication to treat acute pain.

The overall hypothesis is that observational learning influences neural pain modulation and cognition systems, including processes associated with mentalizing (the ability to cognitively understand mental states of others), empathy (the ability to share an emotional experience), and expectancy (the anticipation of a benefit). The objective is to determine the brain mechanisms of observationally-induced analgesia using brain mapping approaches that target changes in blood oxygenation and oscillatory activity in the brain, thus enabling investigators to draw inferences about the localization and extent of neurobiological activation underlying hypoalgesia driven by observation. Therefore, the investigators designed innovative experiments using pharmacological fMRI, EEG, and combined EEG-fMRI measurements.

DETAILED DESCRIPTION:
Analgesic effects can also occur without formal conditioning and direct prior experience because crucial information necessary to build up expectations of analgesia can be acquired through observation of a therapeutic benefit in others. Placebo analgesic effects following the observation of a benefit in another person are similar in magnitude to those induced by directly experiencing an analgesic benefit. These observations emphasize that contextual cues substantially modulate the individual placebo analgesic effects.

In this project, the investigators propose a compelling research agenda to explore the neural mechanisms of hypoalgesia driven by observation as a foundation for future development of novel nonpharmacological pain therapies using pharmacological functional magnetic resonance imaging (fMRI), electroencephalography (EEG), and combined EEG/fMRI. It builds on a decade of experience in placebo research in PI Colloca's lab and with University of Maryland collaborators experienced in brain mapping and pain research. In Aim 1, the investigators will determine the role of endogenous opioids on the neural mechanisms of observationally-induced hypoalgesia by using the opioid antagonist naloxone in a functional Magnetic Resonance Imaging (fMRI) setting. In Aim 2, the investigators will identify the impact of empathy by exploring how being in the immersive environment can enhance observationally-induced analgesia. In Aim 3, the investigators will leverage the EEG/fMRI to determine the neural EEG/fMRI transient changes that could co-occur when socially-induced expectations are violated.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-55 years old)
* English speaker (written and spoken)

Exclusion Criteria:

* Cardiovascular, neurological diseases, pulmonary abnormalities, kidney disease, liver disease, degenerative neuromuscular disease, or history of cancer within past 3 years
* Any history of chronic pain disorder or currently in pain
* Severe psychiatric condition (e.g. schizophrenia, bipolar disorders, mania, autism) and /or psychiatric condition leading to treatment and/or hospitalization within the last 3 years.
* Personal history of mania, schizophrenia, or other psychoses
* Nasal Polyps
* Chronic intranasal drug use ( e.g., intranasal decongestants; antihistamines)
* Lifetime alcohol/drug dependence, or alcohol/drug abuse in past 3 months
* Use of antidepressants, ADHD medication, non-over-the-counter painkillers, methadone, benzodiazepines, barbiturates, and/or narcotics during the past 3 months
* Pregnancy or breast feeding
* Color-blindness
* Impaired, uncorrected hearing
* Left handed
* Allergies or sensitivities to creams, lotions, or food coloring
* Any non-organic implant or any non-removable metal device (e.g., pacemaker, cochlear implants, stents, surgical clips, non-removable piercings)
* Any prior eye injury or the potential of a foreign body in the eye (e.g., worked in metal fields)
* Persistent functional impairment due to a head trauma
* Fear of closed spaces
* Any other contraindications for MRI (e.g., large tattoos on head and neck)
* Previously participated in other "Pain Perception in the Brain" Studies in Colloca lab Failed drug test (testing for opiates, cocaine, methamphetamines, amphetamines, and THC)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neural responses | Two days
  Blood oxygenation level dependent (BOLD) responses will allow the identification of relative activation/deactivation in the brain as result of events (e.g. painful stimulations) that will be given during the experiment and the treatment administration.

SECONDARY OUTCOMES:
Pain ratings | Two days
  Participants will rate painful and non-painful stimulations on a Visual Analogue Scale raging from 0=no pain to 100= maximum unbearable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Luana Colloca, MD/PhD/MS, Principal Investigator — University of Maryland Baltimore School of Nursing
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is neither intent nor plan to share IPD.

REFERENCES:
- [Background] Colloca L. The Placebo Effect in Pain Therapies. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:191-211. doi: 10.1146/annurev-pharmtox-010818-021542. Epub 2018 Sep 14. PMID 30216744
- [Background] Schenk LA, Krimmel SR, Colloca L. Observe to get pain relief: current evidence and potential mechanisms of socially learned pain modulation. Pain. 2017 Nov;158(11):2077-2081. doi: 10.1097/j.pain.0000000000000943. No abstract available. PMID 29035916
- [Background] Benedetti F, Pollo A, Colloca L. Opioid-mediated placebo responses boost pain endurance and physical performance: is it doping in sport competitions? J Neurosci. 2007 Oct 31;27(44):11934-9. doi: 10.1523/JNEUROSCI.3330-07.2007. PMID 17978033